CLINICAL TRIAL: NCT03655886
Title: Cytoreductive Prostatectomy Versus Cytoreductive Prostate Irradiation As a Local Treatment Option for Metastatic Prostate Cancer: a Multicentric Feasibility Trial
Acronym: LoMP II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-01880
Record Dates: First submitted 2018-07-26; First posted 2018-08-31 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer Metastatic
Keywords: metastatic; prostate cancer; local; cytoreductive
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radical prostatectomy (Experimental)
  Interventions: Procedure: radical prostatectomy
- Radiotherapy (Experimental)
  Interventions: Radiation: Whole pelvis radiotherapy

INTERVENTIONS:
Procedure: radical prostatectomy — can be performed either open, laparoscopic or robot-assisted, which is chosen by the discretion and expertise of the performing surgeon
  Arms: Radical prostatectomy
Radiation: Whole pelvis radiotherapy — radiation of prostate bed and pelvis
  Arms: Radiotherapy

SUMMARY:
According to the guidelines of the European Association of Urology (EAU), the first-line treatment for newly diagnosed mPC consists of immediate castration with the addition of docetaxel or abiraterone acetate. As seen in other well-known solid tumours - such as ovarian, colon and renal cancer - local treatment (LT) of the primary tumour could lead to a survival benefit compared to standard of care (SOC). Several retrospective studies have suggested a survival benefit of local treatment of the primary tumour with SOC versus SOC only in mPC. These patients also have less local symptoms of their disease, which has a major impact on quality of life (QoL). Several prospective studies have already been set up to compare either surgery or radiotherapy with the SOC. In expectation of their results and because randomization seems challenging, the investigators want to set up a trial to evaluate the feasibility of randomization between both local treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥18y
* Histologically proven PC
* Newly diagnosed metastatic PC as assessed by standard imaging (CT and bone scintigraphy) or PSMA PET-CT
* ECOG 0-1 (2 if related to local PC symptoms)
* Eligible for local treatment
* Written informed consent and able and willing to comply with protocol requirements

Exclusion Criteria:

* Previous systemic treatment for PC except ADT started within 3 months before randomization
* Previous radiotherapy to the pelvis interfering with prostate irradiation
* Previous surgery in the pelvis interfering with radical prostatectomy
* Symptoms related to metastatic lesions, persisting for at least 2 weeks after initiation of ADT
* Metastatic brain disease, leptomeningeal disease or imminent spinal cord compression
* Previous or current malignant disease which is likely to interfere with LoMP II treatment or assessment
* Psychological disorder intervening with understanding the information or the informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of randomization between both treatment arms as assessed by the randomized proportion | 48 months
  In this trial we want to assess whether it is feasible to randomize patients into both treatment arms. All patients eligible for inclusion will be reported. The eventual proportion of randomized patients will be evaluated. Reasons for exclusion will be monitored.

SECONDARY OUTCOMES:
Radiographic progression-free survival | 48 months
  Calculated starting from date of randomization to radiographic progression or death from any cause whichever occurred first
Clinical progression-free survival | 48 months
  Calculated starting from date of randomization to the date of radiographic progression, symptoms, initiation of new treatment, or death, whichever occurred first.
Quality of life (QLQ-C30 + QLQ-PR25) | 48 months
  Evaluation of quality of life will be done using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire, extended by the QLQ-PR25.
Acute and late toxicity due to local treatment | 48 months
  Early complications after radical prosatatectomy will be evaluated using the Clavien-Dindo classification for surgical complications.
  Acute and late toxicity after radiotherapy will be evaluated using the Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). This outcome will be assessed descriptively, as a direct comparison between the two toxicity classifications would be inappropriate.

OTHER OUTCOMES:
Castration-resistant free survival | 48 months
  Calculated starting from date of randomization until castration-resistant disease development, as defined by the European Association of Urology (EAU) guidelines

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (6):
  - Antwerp University Hospital, Edegem, Antwerp
  - AZ Jan Palfijn, Ghent, East Flanders
  - Leuven University Hospital, Leuven, Flemish Brabant
  - AZ Maria Middelares, Ghent, Ghent
  - AZ Sint-Jan, Bruges, West Flanders
  - University Hospital Ghent, Ghent

IPD SHARING:
Plan to Share IPD: Undecided